CLINICAL TRIAL: NCT00931099
Title: Fetal Outcome of Sleep Disordered Breathing During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Dr. Riva Tauman, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-RT-244-CTIL
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Pregnant Women
Keywords: pregnancy; sleep disordered breathing; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Low risk pregnant women: 300 women in the third trimester of a singleton uncomplicated pregnancy, who attend a low risk obstetric surveillance
- High risk pregnant women: 100 women hospitalized at the Antenatal department due to pregnancy related hypertensive disorder, IUGR, diabetes mellitus or premature labor
- Pregnant women in labor: 200 women of a singleton uncomplicated full term pregnancy will be recruited during labor at the delivery room
- Newborns: 400 newborns belong to women in first two groups

SUMMARY:
Sleep disordered breathing (SDB) is a frequent disorder characterized by some combination of repeated events of partial or complete upper airway obstruction during sleep, disruption of normal ventilation, hypoxemia, and sleep fragmentation. When untreated, SDB is associated with serious cardiovascular and neurobehavioral morbidities. Many physiologic changes that occur during pregnancy may compromise the respiratory system and place women at risk for developing SDB. Indeed, snoring has been reported in up to 46% of pregnant women. Preliminary evidence suggests that SDB is associated with the hypertensive conditions of pregnancy and that oxidative stress and endothelial dysfunction are mechanisms important in the development of both conditions. Moreover, early reports in animals and in humans suggest that maternal SDB may affect the developing fetus and that the intermittent hypoxia and increased sympathetic activity induced by SDB could potentially contribute to adverse maternal-fetal outcome. However, previous reports have focused on crude and non specific measures of fetal outcome such as birth weight and APGAR (Appearance, Pulse, Grimace, Activity, Respiration) score and currently there is no data on the mechanisms underlying the adverse effect of maternal SDB on the fetus and the newborn infant.

Hypothesis: SDB during pregnancy imposes a risk to the developing fetus and the newborn infant through mechanisms mediated by maternal hypoxia.

Objectives:

1. To prospectively investigate the incidence and severity of SDB during pregnancy using an objective tool, i.e., overnight polysomnography (PSG) or at-home sleep study using portable device in a large cohort of pregnant women.
2. To examine the effect of maternal SDB on fetal and neonatal outcome. Methods: 300 women in the third trimester of a singleton uncomplicated pregnancy, who attend a low risk obstetric surveillance will be recruited. Hundred women hospitalized at the Antenatal department due to pregnancy related hypertensive disorder, intrauterine growth restriction (IUGR), diabetes mellitus or premature labor will also be recruited. In addition, 200 women of a singleton uncomplicated pregnancy will be recruited during labor at the delivery room. All participants will be asked to complete a designated sleep questionnaire. Based on the questionnaires, women in the third trimester will undergo a sleep study. Medical records review will be conducted after delivery and will include information of maternal blood pressure, labor duration, route of delivery, infant birth weight and APGAR score. Placentas will be collected immediately after delivery from all women. Cord blood will be obtained immediately after delivery and will be analyzed. Post-natal neurobehavioral evaluation will be conducted. Data analysis will be performed on 4 population subgroups: (1) Sleep study proven SDB, (2) Sleep study proven non-SDB, (3) SDB per questionnaire, (4) non-SDB per questionnaire. Comparisons of fetal outcome measures according to group assignment will be performed. In addition, the association between the severity of SDB based on sleep studies (degree of hypoxemia, degree of sleep fragmentation, amount of respiratory events) and outcome measures will be performed.

DETAILED DESCRIPTION:
Sleep questionnaire: The questionnaire is based on validated questionnaires and includes information on snoring, sleep pauses and daytime sleepiness.Completed questionnaires will be reviewed weekly, and women with either severe daytime sleepiness or self reported frequent snoring or any degree of sleep apnea will be contacted and be requested to undergo clinical evaluation and an overnight polysomnography (estimated - 100 women). This evaluation will consist of an in-depth sleep related and general medical history and physical examination including body mass measurements (height, weight, neck circumference).

Tissue and umbilical cord blood collection: Placentas will be evaluated by a single pathologist. The pathologist will be blind to the medical and perinatal history but not to gestational age. Each placenta will be examined using a criteria previously reported.

Cord blood will be obtained at birth from the double clamped umbilical vein and will be processed immediately for fetal blood gases analysis. Immediately following delivery, 5 mL of blood will be obtained from the umbilical cord of all babies.

Neuro-behavioral evaluation of the newborn will be conducted at the first 48 hours of life.

ELIGIBILITY:
Inclusion Criteria:

* Women in the third trimester of a singleton uncomplicated pregnancy, who attend a low risk obstetric surveillance (for group 1).
* Women with related hypertensive disorder, IUGR, diabetes mellitus, or premature labor (group 2).
* Women of a singleton uncomplicated full term pregnancy at labor (group 3).
* Newborns of women from group 1 and 2 (group 4).

Exclusion Criteria:

* Multiple pregnancies.
* Maternal chronic medical conditions.
* Prematurity.
* Congenital abnormalities.
* Fetal distress.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 300 women in the third trimester of a singleton uncomplicated pregnancy, who attend a low risk obstetric surveillance (group 1). 100 women hospitalized at the Antenatal department due to pregnancy related hypertensive disorder, IUGR, diabetes mellitus, or premature labor will also be recruited (group 2). 200 women of a singleton uncomplicated full term pregnancy will be recruited during labor at the delivery room (group 3). Neonates born to women from group 1 and 2 (group 4).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
neonatal neurobehavioral measures | first 48 h of life, age of 11 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Dunietz GL, Sever O, DeRowe A, Tauman R. Sleep position and breathing in late pregnancy and perinatal outcomes. J Clin Sleep Med. 2020 Jun 15;16(6):955-959. doi: 10.5664/jcsm.8416. PMID 32118576
- [Derived] Kidron D, Bar-Lev Y, Tsarfaty I, Many A, Tauman R. The effect of maternal obstructive sleep apnea on the placenta. Sleep. 2019 Jun 11;42(6):zsz072. doi: 10.1093/sleep/zsz072. PMID 30903184